CLINICAL TRIAL: NCT02462447
Title: Biodistribution and Mechanism of Action of the 11C-labeled PET Tracer Sarcosine in Patients With Prostate Cancer as Well as Radiation Dosimetry, Plasma Pharmacokinetics and Biodistribution in Healthy Volunteers
Brief Title: Carbon-11 Labeled Sarcosine in Prostate Cancer
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Morand Piert, MD, Principal Investigator, University of Michigan
Other Study IDs: HUM00091201; R21CA191052-01 (NIH)
Record Dates: First submitted 2015-02-27; First posted 2015-06-04 (Estimated); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; biopsy; PET
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Group 1 (prostate cancer patients):
  Tissue biopsies from prostate cancer lesions are performed as part of routine clinical care. These tissues will however be used for research purposes.
  Group 2 (healthy men):
  No biopsies are performed in volunteers.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Prostate Cancer: Subjects will receive two PET/CT examinations, one with 11C-sarcosine and one with 11C-choline. These scans will take 30-45 minutes each.
  Interventions: Drug: 11C-sarcosine; Drug: 11C-choline
- Healthy Volunteer: Subjects will receive one PET/CT examination, with 11C-sarcosine. This scan will take approximately 90 minutes.
  Interventions: Drug: 11C-sarcosine

INTERVENTIONS:
Drug: 11C-sarcosine — Radiotracer injection for PET/CT scan
Drug: 11C-choline — Radiotracer injection for PET/CT scan
  Groups: Prostate Cancer

SUMMARY:
Men with and without prostate cancer will have a PET/CT scan that measures the level of the amino acid sarcosine. PET is a scanning method that uses short lived radioactivity.

DETAILED DESCRIPTION:
Tissue levels of the amino acid sarcosine are elevated in prostate cancer compared to normal prostate tissues and further increased in metastases from prostate cancer. This research project is designed to test whether 11C-sarcosine (a chemical that is linked to short lived radioactivity) would be useful to detect prostate cancer in men using PET/CT imaging. The uptake and distribution of 11C-sarcosine in men with known or suspected prostate cancer will be determined and compared with results from 11C-choline PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Males 40 years of age or older
* Confirmed or suspected prostate cancer and will undergo a planned tissue biopsy of the known or suspected tumor (Prostate Cancer Group 1 only)

Exclusion Criteria:

* Active malignancy (except basal cell or squamous cell skin cancer) within the last 2 years
* Body weight > 350 lbs (158 kg)
* Prisoners
* Subject not willing or able to sign informed consent

Min Age: 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: Subjects with confirmed or suspected prostate cancer who will undergo a planned tissue biopsy of the known or suspected tumor
  Group 2: Healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-06; Primary Completion 2017-02-08 (Actual); Study Completion 2017-02-08 (Actual)

PRIMARY OUTCOMES:
Evaluation of biodistribution of 11C-sarcosine in prostate cancer patients | One Month
Evaluation of radiation dosimetry of 11C-sarcosine in healthy volunteers | One Month

SECONDARY OUTCOMES:
Comparison of the uptake measures of 11C-sarcosine with those from 11C-choline | One Month
  Standardized uptake (SUV) values from tumor tissues relative to background, also called tumor-to-background ratios (TBR), will be determined from both, 11C-sarcosine and 11C-choline. Then TBR measurements from 11C-choline and 11C-sarcosine will be compared to identify whether 11C-sarcosine improves tumor to background image contrast relative to 11C-choline in prostate cancer.
Evaluation of underlying metabolic pathways of sarcosine in prostate cancer tissues obtained from tissue materials | One Month
Evaluation of the relationship between sarcosine (and metabolite) tissue concentrations and 11C-sarcosine/11C-choline plasma and tissue uptake measures | One Month

CONTACTS AND LOCATIONS:
Overall Officials: Morand R Piert, MD, Principal Investigator — University of Michigan Hospital
Locations (1):
- University of Michigan Health Systems, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Piert M, Shao X, Raffel D, Davenport MS, Montgomery J, Kunju LP, Hockley BG, Siddiqui J, Scott PJH, Chinnaiyan AM, Rajendiran T. Preclinical Evaluation of 11C-Sarcosine as a Substrate of Proton-Coupled Amino Acid Transporters and First Human Application in Prostate Cancer. J Nucl Med. 2017 Aug;58(8):1216-1223. doi: 10.2967/jnumed.116.173179. Epub 2017 Mar 16. PMID 28302759